CLINICAL TRIAL: NCT02369757
Title: Patients Navigator for Organized Colorectal Cancer Screening in Underserved Population
Brief Title: Patients Navigator for Organized Colorectal Cancer Screening
Acronym: COLONAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); University of Lyon (Other); Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-04
Record Dates: First submitted 2014-12-05; First posted 2015-02-24 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2014-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention of navigators (Experimental): Navigators accompany the target population towards OCCS.
  Interventions: Behavioral: Navigator intervention
- No Intervention (No Intervention): Population is not accompanied by navigators

INTERVENTIONS:
Behavioral: Navigator intervention — peers sharing common characteristics with the target population whose mission is to accompany towards OCCS
  Arms: Intervention of navigators

SUMMARY:
The main objective is to evaluate the impact of the recruitment and training of a peer-navigator on the participation rate of colorectal cancer screening among underserved area. The role of the navigator is to establish an intervention culturally-tailored to the inhabitants in order to promote the Fecal Occult Blood test (FOBT) and accompany the inhabitants to complementary exams, if needed.

ELIGIBILITY:
Inclusion Criteria:

* person living in the IRIS intervention zones
* person invited by the local management structure to participate in colorectal cancer screening

Exclusion Criteria:

* person not living in the IRIS intervention zone
* person not invited by the local management structure to participate to colorectal cancer screening

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40774 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Participation rates | 24 months
  Participation rates between intervention areas and control areas before/after intervention

SECONDARY OUTCOMES:
Percentage of patients primary care peers take care of | 24 months
Qualitative analysis | 1 hour
  A questionnaire will be given to those contacted and some people will be interviewed

CONTACTS AND LOCATIONS:
Overall Officials: Franck Chauvin, PhDMD, Study Chair — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

REFERENCES:
- [Derived] Bourmaud A, Benoist Y, Tinquaut F, Allary C, Ramone-Louis J, Oriol M, Kalecinski J, Dutertre V, Lechopier N, Pommier M, Rousseau S, Dumas A, Amiel P, Regnier V, Buthion V, Chauvin F. Patient navigation for colorectal cancer screening in deprived areas: the COLONAV cluster randomized controlled trial. BMC Cancer. 2023 Jan 6;23(1):21. doi: 10.1186/s12885-022-10169-3. PMID 36609248
- [Derived] Allary C, Bourmaud A, Tinquaut F, Oriol M, Kalecinski J, Dutertre V, Lechopier N, Pommier M, Benoist Y, Rousseau S, Regnier V, Buthion V, Chauvin F. ColoNav: patient navigation for colorectal cancer screening in deprived areas - Study protocol. BMC Cancer. 2016 Jul 7;16:416. doi: 10.1186/s12885-016-2469-9. PMID 27388807